CLINICAL TRIAL: NCT04592263
Title: Patient Centered Care in Diabetes in Ecuador: Mixed-methods Study.
Brief Title: Patient Centered Care in Diabetes in Ecuador
Status: Completed | Type: Observational
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Universidad Catolica Santiago de Guayaquil (Other); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, José Joaquín Mira, Professor, Universidad Miguel Hernandez de Elche
Other Study IDs: CEISH-19-0041
Record Dates: First submitted 2020-10-15; First posted 2020-10-19 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Patient Satisfaction; Patient Engagement; Patient Empowerment; Health Literacy; Patient Experience
Keywords: Patient Reported Measures; Chronic Diseases; Diabetes; Ecuador; Patient Experience; Quality of care
MeSH Terms: conditions — Patient Satisfaction; Patient Participation; Chronic Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Qualitative phase: 4 focus groups and 6 semi-structured interviews.
- Group 2 - Quantitative phase: Pilot study of the tools developed from phase 1.
  Interventions: Other: EPD Questionnaire

INTERVENTIONS:
Other: EPD Questionnaire — A 44 items questionnaire (4 point likert scale) was distributed. Included dimensions where: experience with your physician, provision of care, barriers, outcomes of care, symptoms, patient engagement, health literacy and patient empowerment.
  Other Names: Experience questionnaire of the Person with Diabetes
  Groups: Group 2 - Quantitative phase

SUMMARY:
Introduction: According to World Health Organization data, it is estimated that more than 422 million people have diabetes. In Ecuador, diabetes is the second cause of death, only after ischemic heart disease, and is the first chronic non-communicable disease. The complexity of the pathology, its difficult management and the patient's commitment and involvement in their own care has led health systems to seek mechanisms to activate patients. Currently, tools have been developed, Patient Reported Experience Measures (PREM) and Patient Reported Outcome Measures (PROM), which seek to reduce this gap between patient and health system.

Objectives: To develop and validate PREM and PROM tools for diabetes in the Ecuadorian context. To achieve better clinical results and greater patient satisfaction with the system, thus adding value to the care process of patients with diabetes.

Method: This is a study with two components. The first component will focus on the design and validation of PREM and PROM tools in Ecuador. A second component, consisting of a prospective cohort study for the corresponding implementation of the questionnaires obtained and their validation.

Expected results: It is expected to involve patients in the care process, thus establishing a framework for achieving better clinical outcomes and greater patient satisfaction with the system.

DETAILED DESCRIPTION:
Diabetes is considered a worldwide health problem. Its prevalence is increasing every year despite efforts by health systems in different countries to reduce its impact. Most studies have focused on prevention and the effectiveness of drug treatment and diabetes education. However, in order to achieve greater adherence to therapy we must incorporate one more measure, the activation of patients suffering from this condition. This activation is based, above all, on the perception of self-efficacy, life experience in the face of the disease, confidence that adequate care is being received, and the positive assessment that a better result is being achieved. To achieve this, health systems are committed to redesigning the care process to achieve better short and long term results through the inclusion of patients in the assessment of how the care process is developed (through the patient experience measures) and the results of the care provided (through the outcome measures from the patients' perspective). This approach is being addressed worldwide and is being carried out in various pathologies, such as diabetes and cardiovascular disease, Chronic Obstructive Pulmonary Disease, asthma, etc.

Although the Ecuadorian Health System has undergone a transformation since 2008 with the new constitution and the existing political reform, it has not yet achieved all of its objectives. Despite the significant increase in the number of medical consultations, this is not sufficient as it has not been possible to reflect a real impact on the population. Currently, health systems are aware that it is no longer enough to obtain clinical and administrative data to obtain better clinical results and increase the health of a population, but that they are turning their attention particularly to incorporating the perspective and experience of patients when evaluating the incorporation of changes in the care process. This new focus on patient-centered care is forcing health systems to incorporate new measures to assess the patient's experience through PREMs (Patient Reported Experience Measures) and the results of this care from the patient's perspective through PROMs (Patient Reported Outcome Measure). Thus, at the international level, this type of tool is being developed more and more, and is even being considered in consensus at the international level, a task headed by the International Consortium of Health Outcomes Measures.

In this way, through the development and elaboration, from the perspectives of patients and professionals in the field, tools will be obtained that will allow for adding value to the health care provided by the Ministry of Public Health of Ecuador, expanding the indicators that monitor quality, incorporating patient-centered care and consequently improving clinical results through patient activation and satisfaction.

This is a mixed-methods study. A first component that will focus on the design and validation in Ecuador of PREM and PROM tools through a qualitative study. And a second component, consisting of a prospective cohort study for the implementation of the questionnaires obtained during the first phase that will allow the validation of instruments.

ELIGIBILITY:
Inclusion Criteria:

* Persons with diabetes
* Users of the Health National System
* From rural and urban areas of Ecuador

Exclusion Criteria:

* History of ischemic vascular events. (myocardial infarction and stroke)
* People with neurological or psychiatric pathology that prevents the understanding of the questions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Setting: Primary Care Centers of Ecuador
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcome | 6 months
  Experience questionnaire of the Person with Diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Jose J Mira, PhD, Study Director — Universidad Miguel Hernández de Elche
Locations (3):
- Universidad Católica de Santiago de Guayaquil, Guayaquil, Guayas, Ecuador
- Spain (2):
  - Miguel Hernández University, Elche, Alicante
  - Foundation for the Promotion of Health and Biomedical Research, Sant Joan, Alicante

IPD SHARING:
Plan to Share IPD: Undecided
Available upon reasonable request, and prior consultation with the ethics committee.

REFERENCES:
- [Background] OMS. Informe mundial sobre la Diabetes. Organización Mundial de la Salud. 2016.
- [Background] Mira JJ, Nuno-Solinis R, Guilabert-Mora M, Solas-Gaspar O, Fernandez-Cano P, Gonzalez-Mestre MA, Contel JC, Del Rio-Camara M. Development and Validation of an Instrument for Assessing Patient Experience of Chronic Illness Care. Int J Integr Care. 2016 Aug 31;16(3):13. doi: 10.5334/ijic.2443. PMID 28435422
- [Background] Porter M, Lee TH. The strategy that will fix health care. Harvard Business Review. 2013;94:24.
- [Background] Shah A. Value-based healthcare: A global assessment. Econ Intell Unit. 2016;32
- [Background] Canadian Institute for Health Information. Patient-Centred Measurement and Reporting in Canada Launching the Discussion Toward a Future State. 2017;
- [Background] Ministerio de Salud Publica del Ecuador. Guía de Práctica Clínica (GPC) de Diabetes mellitus tipo 2. 2017;
- [Background] Freire W, Ramirez-Luzuriaga MJ, Belmont P, Mendieta MJ, Silva-Jaramillo K, Romero N, et al. Tomo I: Encuesta Nacional de Salud y Nutrición ENSANUT - ECU 2012. primera ed. Quito: Ministerio de Salud Pública/Instituto Nacional de Estadísticas y Censos; 2014.
- [Background] Barcelo A, Cafiero E, de Boer M, Mesa AE, Lopez MG, Jimenez RA, Esqueda AL, Martinez JA, Holguin EM, Meiners M, Bonfil GM, Ramirez SN, Flores EP, Robles S. Using collaborative learning to improve diabetes care and outcomes: the VIDA project. Prim Care Diabetes. 2010 Oct;4(3):145-53. doi: 10.1016/j.pcd.2010.04.005. Epub 2010 May 15. PMID 20478753
- [Background] Kinmonth AL, Spiegal N, Woodcock A. Developing a training programme in patient-centred consulting for evaluation in a randomised controlled trial; diabetes care from diagnosis in British primary care. Patient Educ Couns. 1996 Oct;29(1):75-86. doi: 10.1016/0738-3991(96)00936-6. PMID 9006224
- [Background] Cinar AB, Schou L. Interrelation between patient satisfaction and patient-provider communication in diabetes management. ScientificWorldJournal. 2014;2014:372671. doi: 10.1155/2014/372671. Epub 2014 Dec 28. PMID 25614885
- [Background] Deshpande PR, Rajan S, Sudeepthi BL, Abdul Nazir CP. Patient-reported outcomes: A new era in clinical research. Perspect Clin Res. 2011 Oct;2(4):137-44. doi: 10.4103/2229-3485.86879. PMID 22145124
- [Background] Mira Solves JJ, Guilabert M, Pérez-Jover V. La medida de la experiencia del paciente en el contexto de una atención centrada en el propio paciente. Rev Española Med Prev y Salud Pública. 2018;XXIII:5-11.
- [Background] Svedbo Engstrom M, Leksell J, Johansson UB, Gudbjornsdottir S. What is important for you? A qualitative interview study of living with diabetes and experiences of diabetes care to establish a basis for a tailored Patient-Reported Outcome Measure for the Swedish National Diabetes Register. BMJ Open. 2016 Mar 24;6(3):e010249. doi: 10.1136/bmjopen-2015-010249. PMID 27013595
- [Background] Prieto Rodriguez MA, March Cerda JC. [Step by step in the design of a focus group-based study]. Aten Primaria. 2002 Apr 15;29(6):366-73. doi: 10.1016/s0212-6567(02)70585-4. No abstract available. Spanish. PMID 11996718